CLINICAL TRIAL: NCT01681290
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of CBX129801 (Ersatta™), Long-Acting Synthetic C-Peptide, in Type 1 Diabetes Mellitus Subjects With Mild to Moderate Diabetic Peripheral Neuropathy
Brief Title: Safety and Efficacy of CBX129801 in Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cebix Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBX129801-DN-201
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Diabetic Peripheral Neuropathy
MeSH Terms: interventions — CBX129801

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CBX129801 High Dose (Experimental): Solution for injection, 2.4 mg, weekly for 52 weeks
  Interventions: Drug: CBX129801
- CBX129801 Low Dose (Experimental): Solution for injection, 0.8 mg, weekly for 52 weeks
  Interventions: Drug: CBX129801
- Placebo (Placebo Comparator): Solution for injection, vehicle with no active, weekly for 52 weeks

INTERVENTIONS:
Drug: CBX129801
  Arms: CBX129801 High Dose; CBX129801 Low Dose

SUMMARY:
The purpose of the study is to determine the beneficial effects of CBX129801 (PEGylated synthetic human C-peptide) following weekly subcutaneous administration for 12 months in type 1 diabetes mellitus patients (T1DM) with mild to moderate diabetic peripheral neuropathy (DPN).

ELIGIBILITY:
Key Inclusion Criteria:

* Give informed consent;
* 18-65 years old;
* Have type 1 diabetes mellitus for a minimum of 5 years, with a stable diabetic regimen (for at least 3 months);
* Have clinical signs of diabetic peripheral neuropathy at screening;
* Have abnormal sural nerve conduction observed bilaterally during screening;
* Be C-peptide deficient;
* Be in good general health (besides having type 1 diabetes mellitus);
* Practice effective contraception during and for at least 12 weeks after study participation;
* Have a body mass index (BMI) ≥18.0 and <35.0 kg/m2.

Key Exclusion Criteria:

* Any significant cardiovascular, hematological, lymphatic, immunologic, urologic, dermatologic, psychiatric, renal, hepatic, pulmonary, endocrine (except for diabetes mellitus), central nervous, gastrointestinal, or other major disease;
* Unstable or inadequate glucose control;
* Any clinically significant laboratory value at screening;
* Occurrence of a severe, unexplainable hypoglycemic event (defined as requiring the assistance of another individual) within 6 months of Day 0, or recurrent episodes of non-severe hypoglycemia (≥3 per week on average) that are deemed clinically significant by the Investigator;
* Have had an islet cell, kidney, and/or pancreas transplant;
* If female, is pregnant or lactating;
* History of alcohol or substance abuse within 2 years;
* Positive screen for hepatitis B, hepatitis C antibody, or human immunodeficiency virus (HIV) antibody;
* Initiation of treatment or change of dose of medication that could affect peripheral nerve function within 60 days;
* Previous treatment with CBX129801 or unmodified C-peptide;
* Receipt of an investigational product or therapeutic device, or participation in a drug research study, within a period of 30 days;
* Chronic use of oral steroids or use of Ampyra (dalfampridine) within 60 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Bilateral change in sensory nerve conduction velocity | Predose and 12 months post dose

SECONDARY OUTCOMES:
Vibration perception threshold | Predose and 6 and 12 months post dose
Clinical composite score | Predose and 6 and 12 months post dose
Pain Intensity due to DPN | Predose and 12 months post dose
Sexual function questionnaires | Predose and 6 and 12 months post dose
Quality of life questionnaire | Predose and 12 months post dose

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Kim, MD — Chief Medical Officer
Locations (28):
- United States (21):
  - Escondido, California
  - Fresno, California
  - Irvine, California
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Torrance, California
  - Tustin, California
  - Walnut Creek, California
  - Atlanta, Georgia
  - Decatur, Georgia
  - Idaho Falls, Idaho
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Butte, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - New York, New York
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
- Canada (2):
  - Toronto, Ontario
  - Laval, Quebec
- Sweden (5):
  - Gothenburg
  - Linköping
  - Malmo
  - Stockholm
  - Umeå

REFERENCES:
- [Derived] Wahren J, Foyt H, Daniels M, Arezzo JC. Long-Acting C-Peptide and Neuropathy in Type 1 Diabetes: A 12-Month Clinical Trial. Diabetes Care. 2016 Apr;39(4):596-602. doi: 10.2337/dc15-2068. Epub 2016 Feb 16. PMID 26884473